CLINICAL TRIAL: NCT02397980
Title: A Multicenter, Randomized Trial to Assess Efficacy of Therapeutic Intervention Programs for Decreasing Caregiver Burden in Caregivers of Patients With Dementia
Brief Title: Intervention Programs for Decreasing Caregiver Burden in Caregivers of Patients With Dementia
Acronym: I-care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Jeong Jee Hyang, Professor, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: EUMC2014-12-028
Record Dates: First submitted 2015-03-13; First posted 2015-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Caregivers
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Basic information about dementia
- Behavioral intervention (Active Comparator): Individual, 90 min a day, with an interval of 2 weeks
  * Education about dementia
  * psychological counselling
  * cognitive behavioral therapy
  Interventions: Behavioral: Behavioral intervention

INTERVENTIONS:
Behavioral: Behavioral intervention — * What the dementia is
  * How to deal with behavioral problems in patients with dementia
  * How to manage caregiver's stress
  * How to care dementic patients as well as caregivers themselves
  Arms: Behavioral intervention

SUMMARY:
The purpose of this study is to investigate if behavioral intervention for dementia caregivers will decrease caregiver burden in caregivers of patients with dementia. This multicenter, randomized trial will be conducted with 80 dementia caregivers, who will be randomized into two groups. One group consists of 40 participants who will receive behavioral intervention and 40 who will not receive intervention (waitlist control). The waitlist control group will be also provided the same intervention after the intervention group has completed the intervention. The behavioral intervention consists of 90-min-session a day with an interval of two weeks for 2 months. The primary outcome measures are the changes in scores of Zaret's Burden Inventory and Philadelphia Geriatric Center for Moral Scale (PGCMS).

DETAILED DESCRIPTION:
This multicenter, randomized trial will be conducted with 80 dementia caregivers, who will be randomized into two groups. One group consists of 40 participants who will receive behavioral intervention and 40 who will not receive intervention (waitlist control). The waitlist control group will be also provided the same intervention after the intervention group has completed the intervention. The behavioral intervention consists of 90-min-session a day with an interval of two weeks for 2 months. The intervention program includes not only the knowledge of dementia and how to manage behavioral problems of patients with dementia but also individual psychological counselling about caregiver's distress. The primary outcome measures are the changes in scores of Zaret's Burden Inventory and Philadelphia Geriatric Center for Moral Scale (PGCMS). Secondary outcomes are changes in scores of neuropsychiatric inventory and Korean -instrumental Activities of Daily Living of patients as well as depression scores of caregivers.

ELIGIBILITY:
Inclusion Criteria:

* 30-80years old
* Caregivers who spend their own time with dementia patients over 4 hours a day
* caregiver distress scores >= 2
* caregivers of patients in Alzheimer's disease dementia ( mild to moderate stage of dementia, Mini-Mental Status Examination:10~26)

Exclusion Criteria:

* illiterate
* severe hearing/visual acuity difficulty
* cognitive impairment

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Caregiver burden (Zaret's Burden Inventory (ZBI) | baseline/10-12 week (after intervention)
  Zaret's Burden Inventory (ZBI)
Changes in quality of life of caregivers as assessed by Philadelphia Geriatric Center for Moral Scale (PGCMS) | baseline/10-12 week (after intervention)
  Philadelphia Geriatric Center for Moral Scale (PGCMS)

SECONDARY OUTCOMES:
Changes in behavioral problems of patients with dementia as assessed by the Neuropsychiatry inventory | baseline/10-12 week (after intervention)
  Neuropsychiatry inventory
Changes in Depression of caregivers as assessed by the geriatric depression scale | baseline/10-12 week (after intervention)
  Geriatric depression scale